CLINICAL TRIAL: NCT01091545
Title: Malmö Breast Tomosynthesis Screening Trial
Acronym: MBTST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Unilabs AB Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 2009/770
Record Dates: First submitted 2010-03-12; First posted 2010-03-24 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; screening; sensitivity; tomosynthesis
MeSH Terms: conditions — Breast Neoplasms; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FFDM+DBT (Other): Single-armed study. Women are their own controls with paired images of digital mammography and breast tomosynthesis.
  Interventions: Radiation: DBT and FFDM

INTERVENTIONS:
Radiation: DBT and FFDM — Women in the study will once undergo both standard FFDM screening (2-views) and DBT (1 view, MLO). This will result in a doubled radiation dose compared to only 2-view FFDM, which is the standard procedure for women in the screening program.

SUMMARY:
To compare digital breast tomosynthesis (DBT) with full field digital mammography (FFDM) regarding effectiveness as screening modalities.

DETAILED DESCRIPTION:
Mammography is the only approved method for breast cancer screening, but not all tumors can be detected with mammography. The main reason is overlapping structures that can either mimic or hide a tumor on a 2-dimensional image like mammography. Digital breast tomosynthesis, (DBT) is a 3-dimensional x-ray technique that has been developed during the last years. A tomographic technique like DBT, which reduces or eliminates the detrimental effect of over- and underlying tissue, can probably help to find more tumors. This study aims to investigate whether more breast cancers can be detected with DBT compared to full field digital mammography (FFDM) in population invited to screening. An interim analysis will be performed during 2013 including the first 7,500 women of the study cohort.

ELIGIBILITY:
Inclusion Criteria:

* women 40-74 years old
* in the regular population based mammographic screening program in Malmö, Sweden.

Exclusion Criteria: pregnancy and women not speaking English or Swedish

-

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for breast cancer detection for DBT and DM respectively | 24 months after trial screening
  Sensitivity and specificity for breast cancer detection will be assessed for DBT and DM respectively. The following screening performance measures will also also investigated: the number of detected cancers per 1000 women screened, the number of recalled women/100 screens (recall rate) after consensus, and the positive predictive value (PPV) for screen-recall and the negative predictive value (NPV), in both reading arms. Analyses of the contribution from different reading steps will be investigated. A follow-up period of 24 months after the intervention period will provide information on the actual numbers of breast cancers in the study population through record linkage with the Swedish Cancer Registry.

SECONDARY OUTCOMES:
What kind of cancers are detected and not detected with DBT? | 24 months after trial screening
  To investigate the biological characteristics of the cancers in the trial by mode of detection (screening detected, interval cancers)
Cost-effectiveness of DBT in screening | 24 months after trial screening
  to investigate the cost-effectiveness of DBT in screening

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Zackrisson, MD PhD, Principal Investigator — Region Skane; Ingvar Andersson, MD PhD, Principal Investigator — Lund University
Locations (1):
- Malmö Breast Screening Unit, Skåne University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Olinder J, Johnson K, Akesson A, Fornvik D, Zackrisson S. Impact of breast density on diagnostic accuracy in digital breast tomosynthesis versus digital mammography: results from a European screening trial. Breast Cancer Res. 2023 Oct 4;25(1):116. doi: 10.1186/s13058-023-01712-6. PMID 37794480
- [Derived] Dahlblom V, Andersson I, Lang K, Tingberg A, Zackrisson S, Dustler M. Artificial Intelligence Detection of Missed Cancers at Digital Mammography That Were Detected at Digital Breast Tomosynthesis. Radiol Artif Intell. 2021 Sep 1;3(6):e200299. doi: 10.1148/ryai.2021200299. eCollection 2021 Nov. PMID 34870215
- [Derived] Zackrisson S, Lang K, Rosso A, Johnson K, Dustler M, Fornvik D, Fornvik H, Sartor H, Timberg P, Tingberg A, Andersson I. One-view breast tomosynthesis versus two-view mammography in the Malmo Breast Tomosynthesis Screening Trial (MBTST): a prospective, population-based, diagnostic accuracy study. Lancet Oncol. 2018 Nov;19(11):1493-1503. doi: 10.1016/S1470-2045(18)30521-7. Epub 2018 Oct 12. PMID 30322817

DOCUMENTS (1):
  • Study Protocol (2009-10-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT01091545/Prot_000.pdf